CLINICAL TRIAL: NCT01961466
Title: Prospective Study on the Influence of Psychosocial Variables (Stress, Type A Behaviour Pattern, Quality of Life of the Diabetic) on Glycemic Balance in Patients With Type 1 and 2 Diabetes.
Brief Title: Diabetes and Psychological Profile
Acronym: DPP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: CHAUVET-GELINIER 2009
Record Dates: First submitted 2013-10-10; First posted 2013-10-11 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Type 1 or 2 Diabetes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetic patients
  Interventions: Other: psychological and social self-administered questionnaires

INTERVENTIONS:
Other: psychological and social self-administered questionnaires

SUMMARY:
This study is based on the analysis of psychological and social questionnaires filled in by diabetic patients whose glycemic balance will be assessed by measuring blood levels of glycated haemoglobin. The aim is to compare glycemic balance by measuring HbA1c in diabetic patients (type 1 and 2) according to whether they have a Type A or B psychosomatic profile evaluated by the Bortner self-questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been given information about the research
* patients with National Health Insurance
* diabetic patients (type 1 or 2)
* patients > 18 ans

Exclusion Criteria:

* Adult patients under guardianship or intellectually dependent
* patients without National Health Insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 or 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Correlations between glycemic balance (HbA1c) and the score on the Bortner self-questionnaire | At 1 year

SECONDARY OUTCOMES:
Scores on the scales | At 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France